CLINICAL TRIAL: NCT01750970
Title: Endoscopic Resection of High Grade(TA, T1, Cis)Non-muscle Invasive Bladder Tumors: Modification of Usual Management of This Resection by Using the Blue Light and Evaluation of the Outcome: Should we Maintain the Dogma of Second Endoscopic Resection as a Principle?
Brief Title: Endoscopic Resection of Bladder Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/34
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Bladder Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resection under blue light (Experimental)
  Interventions: Other: Endoscopic resection under blue light (Hexvix®)
- Resection under white light (Active Comparator)
  Interventions: Other: Endoscopic resection under blue light (Hexvix®)

INTERVENTIONS:
Other: Endoscopic resection under blue light (Hexvix®) — Endoscopic resection

SUMMARY:
To confirm the benefit of endoscopic resection under fluorescence and blue light of high grade non-muscle invasive bladder tumor, and verifying if the second endoscopic resection recommended nowadays can be deleted.

ELIGIBILITY:
Inclusion Criteria:

- 18 year-old and older male and female subjects having high grade non-muscle invasive bladder tumor, with urinary cytology , imaging examination (Ultrasound, urography, or scan) and endoscopic examination

Exclusion Criteria:

- Less than 18 years of age, and having no:

* Non-muscle invasive tumor, and of low grade.
* Bladder tumor infiltrating the muscular layer shown by pre-operative test, with absence of urinary cytology
* No blue light source in sustainable way

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of extra lesions revealed by blue light compared to the resection performed in white light | 2 to 6 weeks after resection

CONTACTS AND LOCATIONS:
Overall Officials: Henry BOTTO, MD, Principal Investigator — Hôpital FOCH 40, rue Worth 92150 Suresnes
Locations (1):
- Hôpital FOCH, Suresnes, France

REFERENCES:
- [Derived] Neuzillet Y, Methorst C, Schneider M, Lebret T, Rouanne M, Radulescu C, Molinie V, Dreyfus JF, Pelcat V, Botto H. Assessment of diagnostic gain with hexaminolevulinate (HAL) in the setting of newly diagnosed non-muscle-invasive bladder cancer with positive results on urine cytology. Urol Oncol. 2014 Nov;32(8):1135-40. doi: 10.1016/j.urolonc.2014.04.005. Epub 2014 Jul 9. PMID 25023786